CLINICAL TRIAL: NCT00590213
Title: An Open Randomised Trial to Compare the Value of Prophylactic Versus Therapeutic Breast Radiotherapy in CASODEX Monotherapy Induced Gynaecomastia and/or Breast Pain in Prostate Cancer Patients
Brief Title: Compare the Value of Prophylactic Versus Therapeutic Breast Radiotherapy in CASODEX
Acronym: COMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, Turkey Clinical Study Information
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7054TR/01
Record Dates: First submitted 2007-12-28; First posted 2008-01-10 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Prostate Cancer
Keywords: Casodex; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Casodex 150mg
Procedure: Radiotherapy
Procedure: Haematology

SUMMARY:
The primary objective of this trial is to examine the value of prophylactic versus therapeutic breast radiotherapy in Casodex monotherapy induced gynaecomastia and/or breast pain. Patients will receive either prophylactic radiotherapy to the breast at a dose of 12Gy (as two fractions of 6 Gy in consecutives days), or will not receive any radiotherapy prior to commencing CASODEX 150mg monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Males patients aged 18 years or over on entry into the trial
* Patients who have non-metastatic cancer that is confirmed by histology or cytology. This primary treatment should have been completed in the last 8 weeks
* The stage should be T1b/T1c/T2/T3/T4 any N category
* Paitents must have given written, fully informed consent to participate in the trial prior to any trial specific assessments being made
* Be able and prepared to comply with trial procedures and restrictions
* Have a life expectancy greater than 2 years

Exclusion Criteria:

* Any known sensitivity to radiation therapy or any conditions which in the investigator's opinion may lead to radiation sensitivity
* Patients with any concurrent malignancy (except for basal cell or TO-2 NO MO squamous cell carcinoma of the skin). History of previous malignancy or treatment for any cancer in the past 5 years
* Previous history of mastectomy including a Webster operation or radiation therapy to the chest area
* Any previous treatment with surgical or medical castration, anti-androgens, monotherapy or oestrogen therapy at any time
* Any evidence of pre-existing gynaecomastia or breast pain
* Patients with history or presence of testicular abnormalities (as CASODEX can potentially aggravate testicular tumours)
* Patients with any concurrent disease or condition that in the opinion of the treating physician, would constitute a hazard for participation in this study or may interfere with the patient's ability to comply with the scheduled visits and assessments. This includes patients whose physical build would prevent reasonable assessment of gynaecomastia
* Liver disease (bilirubin greater than 2.0mg/dL; AST/ALT greater than 2 times the upper limit or normal)
* Patients taking the following drugs; terfenadine, cisapride, astemizole, cyclosporin, and warfarin are excluded from the trial due to the possibility of drug interaction
* Patients with a known history of alcohol abuse
* Concurrent treatment with any druges known to have high potential for causing gynaecomastia or breast pain, eg.Spironolactone, steroid therapy, cimetidine and neuroleptic agents.
* Treatment with a new chemical entity within the previous 4 months or current participation in another clinical trial involving an investigational product
* Patients considered by the investigator to be at risk of transmitting any infection through the body or other body fluids, including acquired immue dificiency syndrome (AIDS) other sexually transmitted diseases or hepatitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2003-06

PRIMARY OUTCOMES:
To examine the value of prophylactic versus therapeutic breast radiotherapy in Casodex monotherapy induced gynaecomastia and/or breast pain

SECONDARY OUTCOMES:
To examine the tolerability of radiotherapy to male breast
To examine the tolerability of Casodex 150mg in localized and locally advanced prostate cancer patients
To examine the efficacy of Casodex 150mg in prostate cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Haluk Ozen, Prof, Principal Investigator — Hacettepe Univ. Med. Fac
Locations (9):
- Turkey (Türkiye) (9):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Diyarbak?r
  - Research Site, Edirne
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Manisa
  - Research Site, Samsun